CLINICAL TRIAL: NCT03393442
Title: Evaluation of Gadolinium Deposits in Healthy Women Participating in a High Risk Screening Program for Early Breast Cancer Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Barbara Bennani-Baiti, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1724/2017
Record Dates: First submitted 2018-01-03; First posted 2018-01-08 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Gd-based Contrast Media Exposure During Breast MRI Scans
Keywords: Magnetic Resonance Imaging; Gd-based contrast media; Gd-deposits; brain imaging; breast cancer screening

STUDY DESIGN:
Intervention Model Description: Female subjects exposed to Gd-based contrast media and female subjects not exposed to Gd-based contrast media will be examined by a diagnostic test (brain MRI scan) to determine the presence or absence of Gd-deposit related signal alterations in the brain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Gd-exposed subjects (Experimental): Diagnostic Test: Brain MRI scan Female subjects at high risk for breast cancer that previously underwent more than 6 Gd-based contrast enhanced MRI exams of the breast.
  Interventions: Diagnostic Test: Brain MRI scan
- 2. Healthy subjects (Active Comparator): Diagnostic Test: Brain MRI scan Age-matched female control subjects that never received Gd-based contrast agents.
  Interventions: Diagnostic Test: Brain MRI scan

INTERVENTIONS:
Diagnostic Test: Brain MRI scan — Diagnostic brain MRI scan with the purpose to detect signal changes due to brain deposits of Gd.

SUMMARY:
Purpose: To determine whether patients at high risk to develop breast cancer having received at least 6 cumulative dosages of macrocyclic Gd-based contrast media in the context of breast cancer screening by means of contrast-enhanced MRI.

Methods: Diagnostic study encompassing two arms: first, 50 patients having received ≥6 dosages of macrocyclic Gd-based contrast media in the course of MRI-based breast cancer screening will undergo brain MRI assessment for signal alterations due to Gd-deposits. The second arm consists of 50 healthy volunteers that never received Gd-based contrast agents, and undergoes the same brain MRI assessment as the patient-based arm 1 of the study. Signal intensities will be compared to assess the potential presence or absence of macrocyclic Gd-based contrast agent deposits in the brain.

In case of presence of signal alterations in arm 1 these will be further stratified by number of previously administered macrocyclic Gd-contrast agent doses.

Projected outcome: High cumulative dosages of macrocyclic Gd-based contrast agent either result or do not result in brain MRI signal alterations in healthy women participating in a high-risk screening program for the early detection of breast cancer that necessitates Gd-contrast agent enhanced breast MRI at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* Female; cumulative exposure to ≥6 dosages of macrocyclic Gd-based agents in the course of breast MRI screening for breast cancer OR no exposure to Gd-based contrast media

Exclusion Criteria:

* Previous chemotherapy; serious illness including cardiovascular and neurological diseases; contraindications to MRI; exposure to non-macrocyclic Gd-based contrast agents

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The examined study population are exclusively female subjects.
Enrollment: 100 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Presence of Gd-deposit associated brain signal alterations | Immediate
  Evaluation of Gadolinium Deposits in Healthy Women Participating in a High Risk Screening Program for Early Breast Cancer Detection in comparison to healthy volunteers without previous Gd-based contrast media exposure - signal intensities of various brain regions measured by different MRI sequences will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Barbara I Bennani-Baiti, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Due to a lack of funding IPD cannot be made publicly available.